CLINICAL TRIAL: NCT00736736
Title: Effects of Hip Abductor and External Rotator Strength Training in Patients With Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200801069R
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-06

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Leg Press (Active Comparator): Leg Press exercise for 3 times/week and sustain for 8 weeks.
  Interventions: Other: Leg Press Exercise
- Hip Exercise (Experimental): Additional hip abductor and hip external rotator strength training to leg press exercise for people in this group. All participants received exercise for 3 times per week for 8 weeks.
  Interventions: Other: Additional Hip Muscle Strengthening to Leg Press Exercise
- Control (No Intervention): Education was given during 8 weeks of study period. After 8 weeks of study, exercise was given as compensation.

INTERVENTIONS:
Other: Additional Hip Muscle Strengthening to Leg Press Exercise
  Arms: Hip Exercise
Other: Leg Press Exercise
  Arms: Leg Press

SUMMARY:
The first purpose was to compare the difference between leg press exercise(LPE) and additional hip abductor and external rotator muscle strength training to leg press exercise(LPE+HAE) in muscle strength, hip kinematics during step down, pain severity and function for patients diagnosed with patellofemoral pain syndrome. The second one was to discover the relationship between the change in muscle strength performance and the difference of hip joint kinematics post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patellofemoral pain syndrome ( Bilateral or unilateral)
* Special tests: crepitus during compression test, patellar grind test (Clarke's sign), pain during compression test, palpation ( at least 2 )
* Below 50 years old
* Pain :after long sitting, up/down stair, squat, kneeling, running & jumping ( at least 2 )
* Pain duration at least 1 month
* At least 1 item of PSS score more than 3 cm

Exclusion Criteria:

* Knee operation
* Central or peripheral neurological deficits
* Obvious knee joint or lower extremity malalignment
* People involved in competitive sports
* PSS sub-scale pain experienced last week more than 8cm
* Have been taking anti-inflammatory drugs , received anti-inflammatory injection or received other therapy for past 3 months

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2008-03; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Muscle Strength by hand-held dynamometry, hip joint kinematics during step down by electromagnetic motion tracking system (FASTRAK, Polhemus ), pain severity by PFPS pain severity scale (PSS), functional performance by Anterior Knee Pain Scale(AKP). | Pre and Post 8 weeks of exercise

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Hwa Jan, Study Chair — The School and Graduate Institute of Physical Therapy of National Taiwan University
Locations (1):
- The School and Graduate Institute of Physical Therapy of National Taiwan University, Taipei, Taiwan

REFERENCES:
- [Background] Mascal CL, Landel R, Powers C. Management of patellofemoral pain targeting hip, pelvis, and trunk muscle function: 2 case reports. J Orthop Sports Phys Ther. 2003 Nov;33(11):647-60. doi: 10.2519/jospt.2003.33.11.647. PMID 14669960